CLINICAL TRIAL: NCT06512896
Title: Clinical Study on the Safety, Tolerability, and Preliminary Efficacy of Intraluminal Injection of FOLactis in Patients With Advanced Solid Tumors Accompanied by Malignant Pleural and Peritoneal Effusion
Brief Title: Clinical Study on Intraluminal Injection of FOLactis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ME-ISV-FOLactis
Record Dates: First submitted 2024-02-08; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2023-08

CONDITIONS: Solid Tumor; Immune Response; Pleural Effusion, Malignant; Peritoneal Effusion
MeSH Terms: conditions — Pleural Effusion, Malignant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The safety and tolerability of intraluminal injection of FOLactis (Other): Evaluate the safety and tolerability of intraluminal injection of FOLactis combined with systemic anti-tumor therapy in patients with advanced solid tumors accompanied by malignant pleural and peritoneal effusion, determine the optimal dose, and explore preliminary efficacy
  Interventions: Other: FOLactis

INTERVENTIONS:
Other: FOLactis — Evaluate the safety,tolerability, efficacy of intraluminal injection of FOLactis combined with chemotherapy, target therapy, and immunotherapy
  Other Names: chemo therapy, target therapy, programmed cell and death protein 1

SUMMARY:
This clinical study is a single arm, prospective, single center clinical study on the safety, tolerability, and preliminary efficacy of a novel FOLactis in situ vaccine in the treatment of advanced solid tumors with malignant pleural and peritoneal effusion. The safety, tolerability and preliminary efficacy of intraluminal injection of FOLactis combined with systemic anti-tumor therapy will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 18 to 80 years old, both male and female;
* Eastern Cooperative Oncology Group Performance Status score 0-2 poinRecurrent or metastatic solid tumors confirmed by pathology (including but not limited to pancreatic cancer, colorectal cancer, lung cancer, liver cancer, cholangiocarcinoma, gastrointestinal stromal tumor, head and neck tumor, gastric cancer, bone and soft tissue sarcoma, neuroendocrine tumor, etc.);
* Malignant pleural/abdominal effusion confirmed by pathology;
* Expected survival time ≥ 12 weeks;
* The main organ function and bone marrow function are normal, meeting the following requirements:

  1. Hemoglobin ≥ 80 g/L (no blood transfusion within 14 days);
  2. Absolute neutrophil count ≥ 1.5 × 109/L, and white blood cell count ≥ 3 × 109/L;
  3. Platelet count ≥ 90 × 109/L;
  4. If there is no liver metastasis, total bilirubin<1.5 × ULN; If there is liver metastasis or Gilbert syndrome in patients with high indirect bilirubinemia, total bilirubin<3 × ULN;
  5. If there is no confirmed liver metastasis, AST and ALT<2.5 × ULN; If there is confirmed liver metastasis, AST and ALT<5 × ULN;
  6. Serum creatinine ≤ 1.5 × The upper limit of normal value (ULN) and the creatinine clearance rate calculated by the Cockroft Fault formula * are ≥ 30 mL/min;
  7. Left ventricular ejection fraction (LVEF) ≥ 50%;
  8. International standardized ratio (INR)<1.5, and activated partial prothrombin time (APTT)<1.5 × ULN.
* The interval between previous anti-tumor therapy and the first administration of this trial is ≥ 4 weeks, and the toxicity related to anti-tumor therapy has returned to ≤ 1 level (excluding hair loss, vitiligo, stable hypothyroidism after hormone replacement therapy, etc.);
* Women of childbearing age must undergo a negative pregnancy test (serum or urine) within 14 days before enrollment, and voluntarily use appropriate methods of contraception during the observation period and within 3 months after the last administration of the study drug; For males, surgical sterilization or agreement to use appropriate methods of contraception during observation and within 3 months after the last administration of the study medication should be considered;
* Those who voluntarily participate and sign an informed consent form, and are willing to follow the experimental treatment plan and visit plan;
* Agree to provide blood samples, pleural/ascitic fluid samples, and histological specimens.

Exclusion Criteria:

* Within 4 weeks prior to enrollment, major surgeries were performed (excluding outpatient minor surgeries such as placement of vascular pathways);
* Even after medication treatment, hypertension is still not well controlled (continuous increase in systolic blood pressure ≥ 150mm Hg or diastolic blood pressure ≥ 100mmHg);
* Suffering from uncontrollable clinical symptoms or diseases of the heart, including: (1) NYHA II and above heart failure; (2) Unstable angina pectoris; (3) Have experienced myocardial infarction within 1 year; (4) Patients with clinically significant supraventricular or ventricular arrhythmias who require clinical intervention;
* Having any history of active autoimmune diseases or autoimmune diseases (such as interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism (which can be included after hormone replacement therapy);
* The patient is currently using immunosuppressive agents or systemic hormone therapy to achieve immunosuppressive effects (dosage>10mg/day prednisone or other therapeutic hormones), and continues to use them within 2 weeks before enrollment;
* Has experienced severe allergic reactions to other monoclonal antibodies; Abnormal coagulation function (INR>2.0, PT>16s), with bleeding tendency or undergoing thrombolytic or anticoagulant treatment, allowing prophylactic use of low-dose aspirin and low molecular weight heparin;
* HIV positive; HCV positive; Uncontrolled active hepatitis B;
* Severe infection (such as requiring intravenous drip of antibiotics, antifungal or antiviral drugs) within 2 weeks before the first medication, or unexplained fever>38.5 ℃ during screening/before the first medication;
* Arterial/venous thrombotic events that occurred within 6 months prior to enrollment, such as cerebrovascular accidents (including temporary ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism;
* Known to be allergic to any investigational drug;
* Pregnant and lactating patients, as well as those with reproductive ability, are unwilling to take effective contraceptive measures;
* Has a clear history of neurological or mental disorders, including epilepsy and dementia;
* Other situations that the researchers believe are not suitable for inclusion. Including but not limited to factors such as family or society, which can affect the safety of the subjects or the collection of data and samples.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | three years
  Evaluate the safety and tolerability of intraluminal injection of FOLactis combined with systemic anti-tumor therapy

SECONDARY OUTCOMES:
Objective Response Rate | three years
  Observation and evaluation of the preliminary efficacy of FOLactis in patients with advanced solid tumors accompanied by malignant pleural and peritoneal effusion
Progression Free Survival | three years
  Changes in the levels of cytokines and lymphocyte subsets in the pleural and peritoneal effusion/peripheral blood of subjects before and after FOLactis treatment;
Overall Survival | three years
  1) The changes in pleural and peritoneal effusion/peripheral blood tumor markers in subjects before and after FOLactis treatment; 2) Changes in tumor microenvironment in the chest and abdominal cavities of subjects before and after FOLactis treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- The Comprehensive Cancer Centre of Nanjing Drum Tower Hospital, Medical School of Nanjing University & Clinical Center Institute of Nanjing University, Nanjing, China, Nanjing, China

IPD SHARING:
Plan to Share IPD: No